CLINICAL TRIAL: NCT00639964
Title: Exploration of the Lipid Metabolism During the Diabetic Pregnancies and Research for New Biological Predictors to Nutritional Interventions
Brief Title: Exploration of the Lipid Metabolism During the Diabetic Pregnancies
Acronym: DIAMANT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Lille (Other)
Collaborators: Ministry of Health, France (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2007/0714; 2007-A00534-49 (Other: ID-RCB number, ANSM); PHRC 2007/R1901 (Other: DHOS); DGS 2007-0340 (Other: AFSSAPS)
Record Dates: First submitted 2008-03-14; First posted 2008-03-20 (Estimated); Last update posted 2025-12-22 (Actual); Status verified 2016-05

CONDITIONS: Pregnancy; Pregnancy in Diabetes; Type 1 Diabetes Mellitus; Type 2 Diabetes Mellitus
Keywords: diabetes; pregnancy; macrosomia; lipidics markers; nutritional factors; placenta; umbilical blood cord
MeSH Terms: conditions — Pregnancy in Diabetics; Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2; Diabetes Mellitus | interventions — Hematologic Tests

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- type 1 diabetic pregnant women (Other): type 1 diabetic pregnant women
  Interventions: Other: blood tests; Other: diet questionnaire; Other: umbilical cord blood collect; Other: placenta collect
- type 2 diabetic pregnant women (Other): type 2 diabetic pregnant women
  Interventions: Other: blood tests; Other: diet questionnaire; Other: umbilical cord blood collect; Other: placenta collect
- healthy pregnant women (Other): healthy pregnant women with normal glucose tolerance
  Interventions: Other: blood tests; Other: diet questionnaire; Other: umbilical cord blood collect; Other: placenta collect

INTERVENTIONS:
Other: blood tests — 3 measures during pregnancy and 1 at post partum, 1 measure at time of delivery from fetal cord
Other: diet questionnaire — questions about nutrition before and during pregnancy
Other: umbilical cord blood collect — collected at the delivery
Other: placenta collect — collected at the delivery

SUMMARY:
Justification:

Intrauterine exposure to type 1 or type 2 diabetes increase the risk of macrosomia (35 % to 50 % versus 10 % in general population) despite a good glycemic control. The consequences are : shoulder's dystocia, lung immaturity, caesarean section, neonatal hypoglycaemia and a high frequency of obesity and metabolic disorders in adults.

The mechanisms of macrosomia are unclear; chronic hyperglycemia and subsequent hyperinsulinaemia observed during the diabetic pregnancy might explain only partially the fetal weight. Considerable interest has been generated over the last decade on the lipids and fatty acids alterations in diabetes pregnancies. Change in lipoproteins metabolism have been described associated with macrosomia. Maternal nutrition before and during pregnancy plays an important role in fetal growth and subsequent development of an increased susceptibility to obesity and diabetes in later life.

Main objective:

Looking for an association between maternal and fetal blood lipid parameters and birth weight and body fat in a context of type 1 or type 2 diabetes.

Secondary objectives:

* Identify lipid markers associated with fetal macrosomia.
* Analyze the placenta by measuring the expression of genes implicated in the storage and the transfer of fatty acids.
* Analyze and compare the expression level of placental genes subjected to parental imprinting and validated in animal models.

DETAILED DESCRIPTION:
Plan of study:

Longitudinal study on 3 groups: 70 type 1 diabetic women, 70 type 2 diabetic women and 70 women with normal glucose tolerance during pregnancy. Recruitment in the department of Diabetology and Obstetrics of CHRU of Amiens and Lille.

Nutritional survey and sampling of blood in the 1st, 2nd and 3rd trimester of pregnancy and at 6 weeks post partum.

Collection of cord blood and placental tissues. Histological and molecular analysis of placenta will be realized both in the departments of Anatomopathology of Lille and Amiens and in Biochemistry Molecular Biology of CHRU of Lille.

Homocysteine and folate assays on cord blood will be centralized in Paris (Hospital St Louis).

Main criteria of judgment

Fetal weight corrected by the gestational age.

Expected results:

* An inverse correlation between maternal and fetal blood fatty acids ratios (polyunsaturated fatty acids/ monounsaturated fatty acids + saturated) and birth weight in the diabetic groups.
* Differences of distribution of fatty acids of maternal and foetal erythrocytic phospholipids correlated with the fetal weight.
* Qualitative and quantitative variations of expression of placental genes such as lipases and genes submitted to parental imprinting.

The biologic parameters will be confronted with the data of the nutritional survey and with glycemic control during pregnancy.

ELIGIBILITY:
Inclusion Criteria:

* pregnant women included before 16 amenorrhea weeks

Exclusion Criteria:

* obesity (BMI > 40kg/m2)
* subject became pregnant with medical infertility treatment
* tobacco > 10
* suspected abuse of alcohol

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 186 (Actual)
Dates: Start 2008-01; Primary Completion 2012-01 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
fetal weight corrected by gestational age | just after delivery

SECONDARY OUTCOMES:
cholesterol (total, HDL, LDL) | 3 measures during pregnancy and 1 at post partum, 1 measure at time of delivery from fetal cord
triglycerides | 3 measures during pregnancy and 1 at post partum, 1 measure at time of delivery from fetal cord
Apolipoprotein A/B rate | 3 measures during pregnancy and 1 at post partum, 1 measure at time of delivery from fetal cord
erythrocytary and plasmatic fatty acid distribution | 3 measures during pregnancy and 1 at post partum, 1 measure at time of delivery from fetal cord

CONTACTS AND LOCATIONS:
Overall Officials: Anne VAMBERGUE, MDPHD, Study Director — University Hospital, Lille; Isabelle FAJARDY, PharmD, Principal Investigator — Univesity Hospital, Lille; Annie MARTIN, PharmD PhD, Principal Investigator — University Hospital, Lille; Gilbert BRIAND, PhD, Principal Investigator — University Hospital, Lille; Jean ROUSSEAUX, MDPhD, Principal Investigator — University Hospital, Lille; Damien SUBTIL, MD, Principal Investigator — University Hospital, Lille; Philippe DUFOUR, MD, Principal Investigator — University Hospital, Lille; Pierre FONTAINE, MDPHD, Principal Investigator — University Hospital, Lille; Philippe DERUELLE, MD, Principal Investigator — University Hospital, Lille; Salha FENDRI, MD, Principal Investigator — Amiens University Hospital; Françoise LE GOUEFF, MD, Principal Investigator — Centre Hospitalier de Roubaix; Delphine VINCENT-DESPLANQUE, MD, Principal Investigator — Centre Hospitalier de Roubaix; Lucie BRESSON, MD, Principal Investigator — Lille University Hospital; Eleonore DELARUE, MD, Principal Investigator — University Hospital of Lille; Odile GAGNEUR, MD, Principal Investigator — University Hospital of Lille
Locations (1):
- CHRU, Lille, Lille, France

REFERENCES:
- [Result] Bouvier D, Rouzaire M, Marceau G, Prat C, Pereira B, Lemarie R, Deruelle P, Fajardy I, Gallot D, Blanchon L, Vambergue A, Sapin V. Aquaporins and Fetal Membranes From Diabetic Parturient Women: Expression Abnormalities and Regulation by Insulin. J Clin Endocrinol Metab. 2015 Oct;100(10):E1270-9. doi: 10.1210/jc.2015-2057. Epub 2015 Jul 24. PMID 26207951